CLINICAL TRIAL: NCT05597332
Title: Effect of Implementing a Care Bundle on the Progression of Acute Kidney Injury in Critical Patients
Brief Title: Care Bundle and Acute Kidney Injury Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Lygia Lussim, Principal Investigator, University of Campinas, Brazil
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 61447422.1.1001.5404
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Care bundle; Critical patients
MeSH Terms: conditions — Acute Kidney Injury | interventions — Patient Care Bundles

STUDY DESIGN:
Intervention Model Description: Before and after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Insertion of care bundle in the electronic medical record of patients who develop AKI.
  Interventions: Other: Care bundle for AKI

INTERVENTIONS:
Other: Care bundle for AKI — To maintain mean arterial pressure (MAP) ≥ 65 mmHg; to keep the patient euvolemic; to avoid nephrotoxic drugs; to adjust dose of medication for kidney function; to exclude urinary obstruction; to monitor urine output and serum creatinine levels.

SUMMARY:
The goal of this clinical interventional study is to learn about the effect of implementing a care bundle in the progression of acute kidney injury (AKI) in critical patients. The main questions it aims to answer are:

* What is the impact of care bundle in AKI progression?
* Some improvement of care bundle adhesion rate through an electronic alert can be achieved?

Participants will be adults and critical patients with AKI. During observational study the incidence and progression of AKI will be measured, as well spontaneous care bundle adhesion by medical team. In the interventional study, the progression rate of AKI influenced by care bundle will be measured, as well the adhesion of care bundle through an electronic alert inserted in the patient's daily medical record.

DETAILED DESCRIPTION:
This is a clinical, multicentric and prospective trial (study type: "before" and "after"). Patients aged ≥18 years, admitted to clinical and surgical intensive care units (ICUs) will be included according to selection criteria.

During observational and interventional studies clinical and laboratorial information from electronic medical records will be registered. AKI diagnosis and classification will be based on serum creatinine levels according to kidney disease improving global outcomes (KDIGO) criteria.

The observational study will be carried out to measure the incidence of AKI KDIGO 1 and its progression rate, in order to estimate sample size for the interventional study. Researchers assumed a 10% to 20% reduction in the progression of AKI KDIGO 1 to more advanced stages after the implementation of the care bundle. In the interventional study, the care bundle will be included in the medical records of each individual who develops AKI KDIGO 1. Patients included in this study will be followed by 7 days from inclusion. Adhesion rate to the care bundle will be measured between observational and interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent ICU admission (≤ 48 hours)
* Patients without AKI or with AKI KDIGO 1 at the time of admission

Exclusion Criteria:

* Patients with chronic kidney disease, stage 4 to 5D
* Patients with kidney transplant
* Patients with AKI KDIGO 2, 3 or on dialysis at the time of inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
AKI progression | ≤ 7 days from inclusion
  AKI progression from KDIGO 1 to KDIGO 2 or 3

SECONDARY OUTCOMES:
Adherence to care bundle | ≤ 7 days from inclusion
  Adhesion rate associated to AKI-care bundle

CONTACTS AND LOCATIONS:
Overall Officials: Lygia Lussim, Principal Investigator — University of Campinas, Brazil

IPD SHARING:
Plan to Share IPD: No